CLINICAL TRIAL: NCT02518555
Title: Early Intervention Trial of Ibrutinib for Patients With Asymptomatic, High-Risk Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Ibrutinib as an Immune Modulating Agent for Patients With Asymptomatic, High-risk CLL/SLL Risk Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Woyach (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Woyach, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-15012; NCI-2015-00932 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-07-09; First posted 2015-08-10 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Diphtheria Toxoid; adacel; Diphtheria-Tetanus-acellular Pertussis Vaccines; ibrutinib; 13-valent pneumococcal vaccine; Influenza Vaccines; fluarix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (concurrent vaccines and ibrutinib) (Experimental): Patients receive ibrutinib PO QD on days 1-28. Patients also receive pneumococcal 13-valent conjugate vaccine IM on day 1 of courses 3 and 5 and trivalent influenza vaccine IM and DTaP vaccine IM on day 1 of course 4. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine Adsorbed; Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Pneumococcal 13-valent Conjugate Vaccine; Other: Quality-of-Life Assessment; Biological: Trivalent Influenza Vaccine
- Arm B (sequential vaccines and ibrutinib) (Experimental): Patients receive pneumococcal 13-valent conjugate vaccine IM on day 1 of courses 1 and 3 and trivalent influenza IM and DTaP vaccine IM on day 1 of course 2. Beginning in course 4, patients receive ibrutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 27 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine Adsorbed; Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Pneumococcal 13-valent Conjugate Vaccine; Other: Quality-of-Life Assessment; Biological: Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine Adsorbed — Given IM
  Other Names: Adacel; Daptacel; Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine; DTaP
Drug: Ibrutinib — Given PO
  Other Names: PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Biological: Pneumococcal 13-valent Conjugate Vaccine — Given IM
  Other Names: PCV13 Vaccine; Prevnar 13
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Trivalent Influenza Vaccine — Given IM
  Other Names: Flu prevention; Flu prophylaxis; Flu shot; Flu vaccination; Fluarix; Fluzone; Influenza Vaccine; Influenza Virus Vaccine, Trivalent, Types A and B; TIV

SUMMARY:
This randomized phase II trial studies how well ibrutinib works when given together with vaccine therapies in treating patients without clinical signs or indications that raise the possibility of a particular disorder or dysfunction (asymptomatic) who have high-risk chronic lymphocytic leukemia or small lymphocytic lymphoma. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Vaccines, such as pneumococcal 13-valent conjugate vaccine, trivalent influenza vaccine, and diphtheria toxoid/tetanus toxoid/acellular pertussis vaccine adsorbed, may help the body build an effective immune response to kill cancer cells. Giving ibrutinib together with vaccine therapies may be a better treatment for chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 2-year progression-free survival of asymptomatic, high-risk genomic chronic lymphocytic leukemia (CLL) patients treated with ibrutinib.

SECONDARY OBJECTIVES:

I. To determine whether concurrent administration of ibrutinib with 2 doses of the pneumococcal vaccine (pneumococcal 13-valent conjugate vaccine) does not negatively impact the immune response compared to those who receive the pneumococcal vaccination with sequential therapy.

II. To determine the safety and toxicity associated with administering ibrutinib to asymptomatic, high-risk genomic CLL patients.

III. To determine the response pattern (complete response [CR] minimal residual disease [MRD]-, CR, partial response [PR], PR with lymphocytosis, stable disease [SD]) in asymptomatic, genomic high-risk patients treated with ibrutinib.

VI. To determine changes in the stress, anxiety and depressive symptoms, and related quality of life indicators from patients treated with ibrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically identified chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) as defined by the World Health Organization (WHO) classification of hematopoietic neoplasms
* CLL/SLL cells must demonstrate one or more of the following high-risk genomic features:

  * Del17p13.1(tumor protein p53 [TP53]) as detected by fluorescence in-situ hybridization (FISH)
  * Del11q22.3 ataxia telangiectasia mutated (ATM) as detected by FISH
  * Complex karyotype (>= 3 cytogenetic abnormalities on stimulated karyotype)
  * Unmutated immunoglobulin variable region heavy chain (IgVH) ( >= 98% sequence homology compared with germline sequence)
  * Zeta-chain (TCR) associated protein kinase 70kDa (ZAP-70) gene promoter hypomethylation < 20%
* No prior therapy for CLL/SLL, including chemotherapy and/or radiotherapy is allowed
* Estimated life expectancy of greater than 24 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Total bilirubin =< 1.5X upper limit of normal (ULN) unless secondary to Gilbert's disease
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5X institutional upper limit of normal
* Serum creatinine =< 2 md/dL or estimated creatinine clearance (CrCl) > 50ml/min/body surface area (BSA)
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time (PTT) (activated partial thromboplastin time [aPTT]) < 1.5 x ULN
* Able to swallow capsules without difficulty and no history of malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or active ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* Female subjects who are of non-reproductive potential (i.e., post-menopausal by history - no menses for >= 1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy); female subjects of childbearing potential must have a negative serum pregnancy test upon study entry
* Male and female subjects who agree to use highly effective methods of birth control (eg, condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], sexual abstinence, or sterilized partner) during the period of therapy and for 30 days after the last dose of study drug

Exclusion Criteria:

* Patients meeting any of the following consensus criteria for initiating treatment for their CLL:

  * Progressive symptomatic splenomegaly and/or lymphadenopathy identified by physical examination
  * Anemia ( < 11g/dL) or thrombocytopenia ( < 100,000/uL) due to bone marrow involvement
  * Presence of unintentional weight loss > 10% over the preceding 6 months
  * National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >= 3 fatigue
  * Fevers > 100.5°F or night sweats for > 2 weeks without evidence of infection
* Patients who have had any treatment for their CLL/SLL, including but not limited to chemotherapy, radiotherapy, or immunotherapy, prior to entering the study
* No corticosteroid use will be permitted within two weeks prior to study, except for maintenance therapy for a non-malignant disease; maintenance therapy dose may not exceed 20 mg/day prednisone or equivalent
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributable to compounds of similar chemical or biologic composition to ibrutinib or any component of pneumococcal, influenza and DTaP vaccines
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject is considered by his or her physician to have a less than 2-year survival expectation
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and/or psychiatric illness/social situations that would limit compliance with study requirements
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization
* Concurrent systemic immunosuppressant therapy (eg, cyclosporine A, tacrolimus, etc., or chronic administration [> 14 days] of > 20mg/day of prednisone) within 14 days of the first dose of study drug
* Patients must discontinue treatment with H2-blockers (cimetidine, ranitidine, etc.) prior to beginning protocol therapy
* Vaccinated with any of the vaccines planned for administration in the trial within 8 weeks of starting treatment on the study
* Recent infection requiring systemic treatment that was completed =< 14 days before starting treatment on the study
* Concomitant use of warfarin or other vitamin K antagonists
* Patients who require treatment with a strong cytochrome P450 (CYP) 3A4/5 inhibitor
* Known bleeding disorders (eg, von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Known history of human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV); patients who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment; those who are PCR positive will be excluded
* Major surgery within 4 weeks of starting trial
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk
* Lactating or pregnant
* Unwilling or unable to participate in all required study evaluations and procedures
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who are alive and progression-free | At 2 years from the date of the first ibrutinib administration

SECONDARY OUTCOMES:
Degree of response (CR MRD-,CR, PR, PR with lymphocytosis, and SD) | Up to 4 years
  Will be summarized across and within cohorts. Will graphically evaluate differences between responders and non-responders in select pharmacodynamic markers across and within arms using side-by-side boxplots. Provided an appropriate number of responses, will fit logistic regression models, with response as the dependent variable, and may find correlations of moderate significance that will merit further research in future studies. Time to treatment failure will be defined as the date of first ibrutinib therapy until the date of next treatment, date of death, or date off-study if due to toxicity, whichever occurs first, censoring patients at last follow-up. Response will be characterized according to a slight modification of the 2008 International Workshop on CLL (IWCLL) guidelines for the diagnosis and treatment of CLL, which include clinical, hematologic, and bone marrow features
Incidence of adverse events, evaluated using the NCI CTCAE version 4.0 | Up to 30 days after study treatment
  In general, the maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed by and across arms to determine toxicity patterns. Toxicity is defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment. The incidence of severe (grade 3+) adverse events or toxicities will be described and reasons patients discontinue study treatment will be summarized.
Proportion of patients who achieve complete response | Within 2 years of starting ibrutinib treatment
  CR requires following for period of at least 2 months while during therapy:
  * Absence of adenopathy, hepatomegaly or splenomegaly on PE
  * Absence constitutional symptoms
  * Normal CBC as exhibited by polymorphonuclear leukocytes ≥ 1500/μL, PLT > 100,000/μL, HGB > 11.0 g/dL (untransfused), and lymphocyte count < 4,000/ μL. Achieve clinical CR lasting for at least 2 months will undergo radiologic eval by CT scans of chest, abd and pelvis. Patients who have radiologic evidence of CR (including absence of lymphadenopathy <1.5cm, absence of hepatomegaly and splenomegaly) will undergo bone marrow aspirate and biopsy
  * Bone marrow aspirate and biopsy must be normocellular for age with <30% of nucleated cells being lymphocytes. Lymphoid nodules absent. Patients who fulfill criteria for CR with exception of having bone marrow lymphoid nodules will be considered a PR
  * 5 color flow cytometry will be used to characterize min. residual dis
Time to next treatment | Date of first ibrutinib therapy until the date of next treatment, assessed up to 4 years
  Will be described across both cohorts by the Kaplan-Meier method.
Time to treatment failure | Date of first ibrutinib therapy until the date of next treatment, date of death, or date off-study if due to toxicity, whichever occurs first, assessed up to 4 years
  Time to treatment failure will be defined as the date of first ibrutinib therapy until the date of next treatment, date of death, or date off-study if due to toxicity, whichever occurs first, censoring patients at last follow-up. Time to treatment failure will be described across both cohorts by the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Woyach, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arrato NA, Valentine TR, Byrd JC, Jones JA, Maddocks KJ, Woyach JA, Andersen BL. Illness representations and psychological outcomes in chronic lymphocytic leukaemia. Br J Health Psychol. 2022 May;27(2):553-570. doi: 10.1111/bjhp.12562. Epub 2021 Oct 4. PMID 34608724
- See also: The Jamesline — http://cancer.osu.edu